CLINICAL TRIAL: NCT04722354
Title: Abscisic Acid Effects on Glucose Homeostasis and Insulin Sensitivity
Acronym: ABA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Collaborators: BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1545505
Record Dates: First submitted 2021-01-08; First posted 2021-01-25 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Pre Diabetes
Keywords: metabolism
MeSH Terms: conditions — Glucose Intolerance | interventions — Abscisic Acid

STUDY DESIGN:
Intervention Model Description: a randomized, cross-over, placebo-controlled trial will be employed to evaluate the effects of ABA (95ug) twice a day (190ug total per day) for 14 days on tolerability and insulin sensitivity during a hyperinsulinemic euglycemic clamp.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABA group (Active Comparator): 95 ug 2x/day for 14 days
  Interventions: Other: Hyperinsulemic euglycemic clamp; Procedure: Muscle Biopsy; Dietary Supplement: Oral abscisic acid (ABA)
- Placebo group (Placebo Comparator): Corn Starch 300 mg for 14 days
  Interventions: Other: Hyperinsulemic euglycemic clamp; Procedure: Muscle Biopsy; Other: Placebo

INTERVENTIONS:
Other: Hyperinsulemic euglycemic clamp — Following a 12-hour overnight fast at the CRU (including abstinence from caffeine containing foods and beverages), insulin sensitivity will be measured using the criterion method of the euglycemic clamp. Participants will have not performed vigorous physical activity for at least the previous 24 h, and be free of acute illness for the prior 2 weeks. An intravenous catheter will be placed in an antecubital vein for subsequent insulin (40 mU/m2-min) and glucose infusions and for stable isotope (6, 6-2H2) infusions to measure insulin sensitivity.
Procedure: Muscle Biopsy — One biopsy taken prior to clamp and a second biopsy taken 30-45 min after the start of the clamp. A biopsy of the Vastus Lateralis muscle will be performed on the leg/thigh using the Bergstrom technique.
Dietary Supplement: Oral abscisic acid (ABA) — Those in this group will receive ABA (95 µg ABA and 300 mg of corn starch)
  Arms: ABA group
Other: Placebo — Those in this group will receive placebo (300 mg cornstarch)
  Arms: Placebo group

SUMMARY:
The purpose of this study is to determine the effects of oral abscisic acid (ABA) on glucose metabolism in subjects with defined prediabetes.

ELIGIBILITY:
Inclusion Criteria

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18-65
4. In good general health as evidenced by medical history or diagnosed with <specify condition/disease> or exhibiting <specify clinical signs or symptoms or physical/oral examination findings>
5. Fasting glucose >5.6 and<7.0 mmol/L and/or HbA1C >5.6 and <6.5 %
6. Ability to take oral medication and be willing to adhere to the <study intervention> regimen
7. Females currently on hormone replacement therapy (HRT) can participate in the study if they have been on HRT for at least 6 months and will continue to be on HRT during the study.
8. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner
9. Agreement to adhere to Lifestyle Considerations throughout study duration.

Exclusion Criteria

1. Treated or untreated diabetes
2. 19>BMI<40.0 kg/m2
3. Blood pressure (BP) ≤ 150mmHg systolic and ≤ 95 mmHg diastolic
4. Current use of medications or antioxidant vitamins or supplements that would impact dependent variables, including glucose metabolism.
5. Past or current ischemic heart disease, stroke, respiratory disease, endocrine or metabolic disease, neurological disease, hematological-oncological disease and free of recent infection (prior 2 weeks)
6. Pregnancy or lactation
7. Treatment with another investigational drug or other intervention within 1 year.
8. Current smoker or tobacco use within the past year.
9. Disqualifying findings on physical examination include cardiac murmurs, diminished pulses or the presence of bruits in the lower extremities, lower extremity thrombophlebitis, evidence of peripheral neuropathy, paresis or edema.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Monitoring adverse events | 10 weeks
  Adverse events will be monitored at each visit throughout the duration of the study.
Insulin sensitivity | 4-6 hours
  Insulin sensitivity will be measured using hyperinsulinic euglycemic clamp

CONTACTS AND LOCATIONS:
Overall Officials: Bret Goodpaster, PhD, Principal Investigator — Principal Investigator
Locations (1):
- AdventHealth Translational Research Institute, Orlando, Florida, United States